CLINICAL TRIAL: NCT01349634
Title: A Study to Measure the Effect of Switching the Salt Supply From Non-iodized to Iodized on Cognitive Development in Ethiopia
Brief Title: The Effects of Iodized Salt on Cognitive Development in Ethiopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Micronutrient Initiative (Other); Ethiopian Health and Nutrition Research Institute (Other)
Responsible Party: Principal Investigator, Grace S. Marquis, Associate Professor, Canadian Research Chair in Social and Environmental Aspects of Nutrition, McGill University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10-1152-MCGUNI-01
Record Dates: First submitted 2011-04-20; First posted 2011-05-06 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Iodine Deficiency; Goiter; Cretinism
Keywords: iodine; goiter; cretinism; child nutrition; cognition
MeSH Terms: conditions — Goiter; Congenital Hypothyroidism | interventions — iodized salt

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Comparison group (No Intervention): This arm will use the salt that is on the open market, which is primarily non-iodized salt. Iodized salt may enter in these communities through the normal trade route. No active interference with salt trade will occur in these communities.
- Early delivery of iodized salt (Experimental): Iodized salt that is produced nationally for the open market (which meets only about 10% of national needs) will be directed to these communities through the normal trade system or by direct delivery to the communities.
  Interventions: Other: Iodized salt

INTERVENTIONS:
Other: Iodized salt — salt for human consumption is fortified at the national level with iodine. The experimental group will receive iodized salt early. the comparison group will receive it by market forces. presently there is only enough iodized salt to meet 10% of the countries needs, and is targeted mainly to urban areas.
  Arms: Early delivery of iodized salt

SUMMARY:
Many school children in Ethiopia and their mothers are known to be iodine deficient. Prevalence in the Amhara region is around 29%. Micronutrient Initiative, a development organization based in Ottawa, plans to help iodize the salt by providing iodization machines and iodine to the salt producers in Lake Afdira where salt is produced and distributed to the population of Ethiopia. Although it is generally assumed that iodine is important for cognitive development, very few studies examining the effects of iodized salt have been conducted. Studies using a single dose of iodine capsules with children 6 to 12 years showed mixed outcomes with approximately 25% yielding positive outcomes for the intervention children. Sixty districts in Amhara will be randomly selected and randomly assigned so that half receive early delivery of iodized salt. Approximately 6200 mothers and their children 6-, 18-, or 60-months old will be recruited from 1-2 villages in each of the 60 districts, with the help of government-paid Health Extension Workers, for a 12-mo longitudinal study starting in May 2011, prior to the introduction of iodized salt. These same mothers and children will be visited 12 months later for repeated measures. Measures include nutritional status such as height and hemoglobin, along with iodine sufficiency (e.g., goitre, urinary iodine, thyroglobulin), and child development (Bayley Scales of Infant and Toddler Development III, Wechsler Preschool and Primary School Intelligence test for older children). Comparisons will be made within and between groups to determine whether iodized salt has an effect on children's mental development.

DETAILED DESCRIPTION:
MATERIALS AND METHODS Sample size was estimated on the basis of the Bayley Scales of Infant and Toddler Development III (Bayley) where the mean is 100 and the standard deviation is 15. Using an effect size of 0.20 standard deviation, a beta of .05 and power of .80, and accommodating for clustering within villages and attrition, the investigators require a sample size of 800 for each group (intervention and control). Severely anemic children (< 8 mg/L) will be referred for treatment and not included in the study.

In this longitudinal study the investigators will recruit 3200 6-mo old infants and 1600 children from each of two other age groups: 18-, and 60-months (inclusion criteria) and their mothers. The exclusion criteria: severe anemia (hemoglobin < 8g/dL). If children are too disabled to take a cognitive test, this will be noted but no cognitive testing administered.

From six zones around Bahir Dar, the investigators will randomly select 60 districts. Half will be assigned randomly to start receiving iodized salt in July 2011; the other half will receive iodized salt as it becomes available in the market. From each district, 1-2 villages will be randomly selected for recruiting 30 children from each age group. It is assumed that with a pregnancy rate of 3.7%, approximately 166 children are born every year in a village of 4500, and 13 are born every month. So within 3 months, starting in May 2011, 30 children of each age could be recruited.

With the help of Health Extension Workers, trained field workers will identify the participants : children of eligible age. Mothers will provide written consent for themselves and their children to participate.

Mothers will be interviewed at baseline and endline concerning the family's economic and demographic information, child's health and diet, and opportunities for stimulation of children (Home Observation for Measurement of the Environment Inventory; Center for Epidemiologic Studies Depression Scale symptom scores). Children's nutritional status will be measured with a food frequency questionnaire, length/height, weight, blood indicators for thyroid function (thyroglobulin, thyroxin, triiodothyronine) and iron status (hemoglobin, ferritin, soluble transferrin receptor), and inflammation (C-reactive protein), goiter, and urinary iodine. A maximum of 10 mL will be collected for blood by venipuncture. Finally, trained assistants will administer the Bayley Scales of Infant and Toddler Development III (cognitive, language, and fine motor scales) to children under-3 years and two Wechsler Preschool and Primary School Intelligence test subscales and School Readiness test for 60-month olds. Salt will be collected at various places of purchase and in households to test for iodine content (first qualitatively, then quantitatively if iodized) at baseline and at the end of the study. All data collection will be done at home or a convenient site in the village.

Conversion of diet into iodine content will be done based on food composition table. Anthropometric data will be converted to standardized scores using the new World Health Organization reference curves, using World Health Organization's software Anthro v. 2 for children up to 60 months of age.

Analyses will compare the nutritional and developmental outcomes of two groups who differ in iodized salt exposure, covarying confounders such as mother's education, family assets, child's sex, and adjusting for clustering. Developmental scores will be derived for the Bayley subtests, and the Wechsler Preschool and Primary School Intelligence test. These tests typically assign 1 point for every correct answer and 0 points for incorrect answers; the summed continuous scores are then used for analysis. Potential confounds include the Home Observation for Measurement of the Environment Inventory and Center for Epidemiologic Studies Depression Scale symptom scores, which also are calculated as the sum of individual item points. Laboratory analyses will be conducted to determine hemoglobin, ferritin, soluble transferrin receptor, thyroglobulin, thyroxin, and triiodothyronine from blood samples, and iodine excretion from urine samples. Analyses of salt will also indicate whether salt consumed by participants in the intervention districts has the required ppm of iodine and more than salt consumed in control districts. If households in the control sites have higher than expected levels of iodine, this will be recorded and included in the analyses.

ELIGIBILITY:
Inclusion Criteria:

* children within 15 days of 6, 18, and 60 months

Exclusion Criteria:

* severe cognitive impairment so child cannot respond to Bayley Scales of Infant and Toddler Development III test

Ages: 5 Months to 61 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5704 (Actual)
Dates: Start 2011-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
cognitive development at 6 mo | 6 months
  Bayley Scales of Infant and Toddler Development III cognitive, language, and fine motor scales
Cognitive development at 18 mo | 18 months
  Bayley Scales of Infant and Toddler Development III cognitive, language, and fine motor scales
cognitive development at 60 mo | 60 months
  two Wechsler Preschool and Primary School Intelligence subscales plus a School Readiness test

SECONDARY OUTCOMES:
nutritional status at 6 mo | 6 months
  weight, length/height, iodine and iron status
nutritional status at 18 mo | 18 months
  weight, length/height, iodine and iron status
nutritional status at 60 mo | 60 months
  weight, length/height, iodine and iron status

CONTACTS AND LOCATIONS:
Overall Officials: Grace S Marquis, PhD, Principal Investigator — McGill University; Frances Aboud, PhD, Principal Investigator — McGill University; Aregash Samuel, MSc, Principal Investigator — Ethiopian Health and Nutrition Research Institute
Locations (1):
- McGill University, Montreal, Quebec, Canada